CLINICAL TRIAL: NCT07319221
Title: Accuracy of Artificial Intelligence Technology in Detecting Number of Root Canal of Human Mandibular Second Molar: Diagnostic Accuracy Experimental Study
Acronym: AI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Amr Mortada Tony AL-Hadary, B.D.S Dental College, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: FUE.REC (46)/11-2024
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Detecting Number of Root Canal of Human Mandibular Second Molar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- morphology of canals in lower second mandibular molar (Experimental): Anatomical variations in root canal systems, such as the presence of an additional root canal, are common, and failure to detect all canals can lead to treatment failure.
  Interventions: Procedure: CBCT
- Number of canals in lower second mandibular molar (Experimental): Number of canals in lower second mandibular molar
  Interventions: Procedure: AI

INTERVENTIONS:
Procedure: AI — Detection of all canals in patients indicated for root canal therapy in lower second molars by Artificial Intelligence Dental operating microscope and CBCT
  Arms: Number of canals in lower second mandibular molar
Procedure: CBCT — CBCT scans performed to all participants, will be randomly distributed upon postgraduate students using randomization software
  Arms: morphology of canals in lower second mandibular molar

SUMMARY:
to detect the Accuracy of Artificial Intelligence Technology in Detecting Number of Root Canal of Human Mandibular Second Molar: Diagnostic Accuracy Experimental Study.

ELIGIBILITY:
Inclusion Criteria:

-

A- Inclusion criteria:

1. Patients must be medically free from any systemic disease that can affect root canal treatment.
2. Age range of the patients should be 18-40 with permanent mandibular second molars indicated for root canal treatment.
3. No sex predilection.
4. Patients must have good oral hygiene.
5. restorable teeth.
6. Positive patient"s acceptance for participating in the study.
7. Patients able to sign informed consent.

B- Exclusion criteria:

1. Lower second molars which are non-restorable, having large perforations, external root resorption, vertical root fracture, internal root resorption, grade 2/3 mobility, previous successful/non-successful root canal treatment
2. Pregnant women after taking detailed history and pregnancy test must be in the first visit.
3. Psychologically disturbed patients.

   Teeth that have:

   • Periodontally affected with grade 2 or 3 mobility. 12

   • Not restorable teeth.

   • Abnormal anatomy and calcified canals.

   • Previous root canal treatment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-11-29 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Number of root canals detected | within one year
  Detected by AI software

CONTACTS AND LOCATIONS:
Locations (1):
- Future University Dental Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: with in one year